CLINICAL TRIAL: NCT01167348
Title: The Effectiveness Of Auricular Acupressure On Body Weight Parameters On Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TsaoTun Psychiatric Center, Department of Health, Taiwan (Other)
Responsible Party: Han-Yi Ching, Psaotun psychiatric center,department of health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tsaotun Psychiatric Center
Record Dates: First submitted 2010-07-16; First posted 2010-07-22 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Schizophrenia; Obesity
Keywords: auricular acupressure; obesity; schizophrenia; body weight
MeSH Terms: conditions — Schizophrenia; Obesity; Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: auricular acupressure — Investigator will put a tape with a 0.5mmx0.5mm seed on the specific positions on the ear of participants of intervention group, and participants will be asked to press these specific positions 3 times a day.

SUMMARY:
The purpose of this study is to examine whether auricular acupressure is effective in reducing body weight, waist circumference, or lipid profile.

ELIGIBILITY:
Inclusion Criteria:

1. ICD:295,living in chronic ward for more than 2 month
2. Body Mass Index (BMI) >or=24
3. Age between 20 to 60
4. Psychotic status stable and can communicate

Exclusion Criteria:

1. Unstable psychotic status
2. Participants who have endocrine disease
3. Participants who have cardiac disease
4. Participants who have immunological disease
5. Participants who have liver or renal function impairment
6. Pregnant woman or in milking stage
7. Cerebrovascular accident (CVA) stroke and disability
8. Participant who attends weight control programs in recent 3 months
9. Any conditions that clinical doctors refuse to let join in this study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Using Body weight scale (kilogram) and checking body weight for all participants | 2 months
  all participants are going to be measured body weight per week for 2 months.

SECONDARY OUTCOMES:
waist circumference | 2 months
  All participants are going to be measured waist circumference per week for 2 months.
Fat percentage by using bio-Impedance Analysis(Tanita-519 machine) | 2 months
  All participants will be measured fat percentage by BIA(Tanita-519) per 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ching Han-Yi, MD, Principal Investigator — Tsaotun Psychiatric Center
Locations (1):
- Tsao-Tun Psychiatric Center, Nantou City, Taiwan